CLINICAL TRIAL: NCT03693911
Title: ACT to Prevent Eating Disorders: Evaluation of the AcceptME Digital Gamified Prevention Program Based on Acceptance and Commitment Therapy
Brief Title: ACT to Prevent Eating Disorders: Evaluating a Gamified Prevention Program
Acronym: AcceptME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Maria Karekla, Assistant Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ΕΕΒΚ/ΕΠ/2013/05-2
Record Dates: First submitted 2018-09-30; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: High Risk for Eating Disorder; Eating Disorders in Adolescence; Acceptance Processes
Keywords: gamification; Acceptance and Commitment Therapy; digitalized intervention
MeSH Terms: conditions — Behavior | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Comparison between AcceptME and waitlist control group
Masking Description: No masking was carried out
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention group (Experimental): AcceptME- digital gamified Acceptance and Commitment Therapy prevention program
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Waitlist control (No Intervention): Waitlist control group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — 6 digital and gamified session prevention program based on Acceptance and Commitment Therapy
  Other Names: AcceptME
  Arms: Prevention group

SUMMARY:
Eating Disorders (ED) constitute a serious public health issue that affects predominantly women and appears typically in adolescence or early adulthood. ED are extremely difficult to treat as these disorders are ego-syntonic and many patients do not seek treatment. As ED are associated with significant adverse medical and psychological consequences, it is vital to focus on the development of successful prevention programs. Even though, in the last two decades significant steps have been made over the development of efficacious and effective ED prevention programs, there is room for improvement in regards to effect sizes. Prevention programs for ED to date have focussed on either reducing the pursuit of the thin ideal or on disputing and replacing unrealistic thoughts with regard to food, body and weigh. There is a growing body of evidence supporting the functional relationship between ED symptomatology and control of emotional states either by avoiding or inhibiting emotional responses. The present study aimed to investigate the effectiveness and acceptability of a digital Acceptance and Commitment Therapy (ACT) based prevention program in comparison to a wait-list control group for young women identified to be at risk for ED. The goals of the study were to describe the development of the AcceptME protocol and digitalized program, assess participants' feedback and the acceptability of the program, and examine the effectiveness of the ACT-based prevention program compared to a wait-list control group. This prevention program has several innovations: a) it is based on ACT theory and practices; b) it uses gamification principles to create a program appealing to adolescents; c) it targets behaviour change in individuals via helping a digital character overcome difficulties in the digitalized program.

DETAILED DESCRIPTION:
Eating Disorders (EDs) constitute a serious public health issue that affects mainly women and appears typically in adolescence or early adulthood. EDs often result in serious physical health consequences as well as enduring psychological difficulties and behavioral complications. Prevention of EDs is paramount as it will reduce such adverse effects, improve the quality of the patient's and his/her family's life and decrease costs incurred by EDs. To date, prevention approaches have not been uniformly effective for EDs and as a consequence there is great room for improvement. There is a growing body of evidence supporting the functional relationship between EDs symptomatology and controlling emotional states either by avoiding or inhibiting the emotional response. Furthermore, theories support that AN begins with a general need of self control and not just emotional control. Current prevention programs for EDs have largely ignored on the problem concerning self-control. This study will propose a new prevention program based on the cognitive-behavioral theory, which suggests that one of the main features of anorexia is a general need of self-control, and the psychological inflexibility theory, which suggests that this need of experiential control may lead to a broader state of psychological inflexibility. A prevention program based on mindfulness, acceptance and change is hypothesized to be able to target ineffective control strategies in individuals at high-risk for developing EDs, prior to the disorder manifesting itself. A treatment which is based on mindfulness and acceptance is Acceptance and Commitment Therapy (ACT), a 3rd wave CBT that targets ineffective control strategies and inflexibility found in a range of psychopathology problems. This study will apply an ACT based prevention program for EDs in an internet based delivery modality delivered to high-risk individuals. The hypotheses made are the following: participants receiving the prevention program will 1) develop greater body image flexibility, 2) decrease their control behaviours (e.g. dieting, exercising, body image avoidance behaviors), and 3) have significantly fewer ED symptoms, decreased body dissatisfaction, decreased risk for developing EDs and have significantly higher quality of life, as compared to the wait-list control group at the end of prevention and at 1-month follow up. We also hypothesized that changes in ACT-related process measures (defusion, mindfulness, values, willingness, body image flexibility, self as context) will mediate improvements in EDs outcome measures (eating disorder risk, eating disorder symptoms, dieting, exercising, body image avoidance behaviour). For the purposes of the study, high-risk participants developing EDs will be recruited from high schools and vocational schools. Participants will be randomly assigned either to the internet-based ACT intervention or the wait list control group. Participants will complete process and outcome measures at baseline, post treatment and follow-up. Results will be then analyzed and conclusions will be made. Repeated measures MANOVA will be used to assess the changes and the differences between the prevention group and the wait list control group. Furthermore, to assess whether ACT variables such as values, mindfulness, defusion, self as context, willingness will mediate ED symptoms mediation analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* females
* aged 13-25 years,
* voluntary participation and parental consent for ages lower than 18 years,
* good working knowledge of the Greek language and
* report a score of greater that 52 at the Weight Concern Scale (Killen et al., 1996) thus, indicating that they are at high risk for developing ED.

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 92 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Risk for developing an Eating Disorder | Post-intervention (following completion of digital session 6, approximately 6 weeks) and follow-up (1 month after post-intervention, approximately 10 weeks)
  Change in risk for developing an Eating Disorder as assessed via the Weight Concerns Scale (WCS; Killen et al., 1994) assessing fear of weight gain, worry about weight and body shape, the importance of weight, diet history, and perceived fatness. Specifically, scores above 52 are associated with an increased risk of developing an eating disorder within 4 years for adolescent girls (Killen et al.,1996).
Body Image Inflexibility | Post-intervention (following completion of digital session 6, approximately 6 weeks) and follow-up (1 month after post-intervention, approximately 10 weeks)
  Change in Body Image Inflexibility as assessed via the Body Image-Acceptance and Action Questionnaire (BI-AAQ; Sandoz et al., 2009). This scale assesses body image acceptance, "the extent to which an individual actively contacts perceptions, thoughts, beliefs, and feelings about his or her body without directly attempting to change their intensity, frequency or form" (Sandoz et al., 2009, p. 8). Scores range from 7-84. Higher summed scores indicate higher body image inflexibility.

SECONDARY OUTCOMES:
Body Dissatisfaction | Post-intervention (following completion of digital session 6, approximately 6 weeks) and follow-up (1 month after post-intervention, approximately 10 weeks)
  Change in Body Dissatisfaction as assessed via the Body Shape Questionnaire-8C (BSQ-8C; Cooper et al., 1987). is a self report short version of the 34-item BSQ, assesing body dissatisfaction as a result of feelings of being fat. The BSQ-8C includes 8 questions extracted from the full version and it was found to be the most favorable version according to Pook and colleaques (2008), as it presented with excellent treatment sensitivity to change in the course of therapy. It is rated on a 6-point scale from "never" to "always. Higher scores indicate more body dissatisfaction.
Quality of life | Post-intervention (following completion of digital session 6, approximately 6 weeks) and follow-up (1 month after post-intervention, )approximately 10 weeks
  Change in Quality of life as assessed via the Youth Quality of Life Instrument-Short Form (YQOL-SF; Patrick & Edwards, 2013). The short-form includes 15 questions assessing domains of sense of self, social relationships, environment and general quality of life. The response scale ranges from 0 (not at all) to 10 (completely). The scores are summed and then transformed to a 0 to 100 scale, with a higher score representing higher quality of life.
Eating Disorder Symptomatology | Post-intervention (following completion of digital session 6, approximately 6 weeks) and follow-up (1 month after post-intervention, approximately 10 weeks)
  Change in Eating Disorder Symptomatology as assessed via the Eating Disorder Examination Questionnaire (EDE-Q; Fairburn & Beglin, 1994). It is a self report version of the EDE interview, assessing the frequency of key behavioural features of eating disorders (i.e., measures the number of times and days a behaviour has occurred in a 4-weeks period). Four subscales (Restraint, Weight Concern, Shape Concern and Eating Concerns) and a global score is derived. The global score is used for purposes of this study.

OTHER OUTCOMES:
Cognitive Defusion | Assessed at the beginning of each of the 6 digital sessions
  Change in Cognitive Defusion as assessed via the Figurative Cognitive Fusion Scale (FCDS; Karekla & Nikolaou, 2011). This is a single item scale assessing cognitive fusion schematically by indicating the relation between ones' self and worrisome thoughts (e.g. regarding body weight and shape in this case). The scale range is 1-10 with higher scores indicating greater levels of cognitive defusion whereas lower scores indicating more cognitive fusion.
Values consistent actions | Assessed at the beginning of each of the 6 digital sessions
  Change in Values consistent actions as assessed via the The BULLs-eye Instrument of valued life (Lundgren & Dahl, 2006). This is a self report instrument evaluating participants' level of consistency and persistence in living in accordance to their values (rated on a scale from 1-10). The domains of value living are friendships/family, education/work, relationships/dating and health. Scores on each domain are averaged to yield an overall score. Higher scores indicate greater consistency in pursuing valued activities.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Karekla, PhD, Principal Investigator — University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Non-US/Non-Canadian, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided